CLINICAL TRIAL: NCT04869800
Title: A Randomized, Open-label, Single Dose, Crossover Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-398 in Healthy Volunteers Under Fasting Conditions
Brief Title: Evaluate the Drug-drugs Interaction Between Lobeglitazone 0.5mg and Empagliflozin 25mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A113_01BE2103
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): 1. Period 1: Reference drug(CKD-501, D745)
  2. Period 2: Test drug(CKD-398)
  Interventions: Drug: CKD-398; Drug: CKD-501, D745
- Sequence 2 (Experimental): 1. Period 1: Test drug(CKD-398)
  2. Period 2: Reference drug(CKD-501, D745)
  Interventions: Drug: CKD-398; Drug: CKD-501, D745

INTERVENTIONS:
Drug: CKD-398 — Test Drug
Drug: CKD-501, D745 — Reference Drug

SUMMARY:
A Clinical Trial to evaluate the Pharmacokinetics and Tolerability of CKD-398

DETAILED DESCRIPTION:
A randomized, open-label, single dose, crossover study to evaluate the pharmacokinetic profiles and safety of CKD-398 in healthy volunteers under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults age≥19 years and age<55 years at the time of screening
2. Individuals who had 17.5 kg/m2 ≤ Body Mass Index(BMI) < 30.5kg/m2 and men's total body weight ≥ 55 kg, women's total body weight ≥ 45 kg

   * BMI = Weight(kg)/ Height(m)2
3. Individuals without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination within the last 3 years
4. Individuals who were deemed to be appropriate as study subjects following laboratory tests (hematology, blood chemistry, urinalysis, viral/ bacterial, etc.) and vital signs, ECG etc. performed at screening
5. Individuals who signed an informed consent form approved by the IRB of Chonbuk National University Hospital and decided to participate in the study after being fully informed of the study prior to participation, including the objective, content and characteristics of the investigational product
6. Individuals who agreed proper contraception during the study and did consent to not donation of sperm 1 month after the last dose of study drug infusion
7. Individuals with the ability and willingness to participate the entire study period

Exclusion Criteria:

1. Individuals with a medical evidence or a history (excluding a dental history of periodontal surgery, impacted wisdom teeth removal, etc.) of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurologic or immune diseases.
2. Individuals with a medical history of gastrointestinal disease (e.g., gullet disease such as esophageal achalasia and esophagostenosis and Crohn's disease) or operations (excluding simple appendectomy, herniotomy or tooth extraction) that may affect drug absorption.
3. Individuals with the following laboratory test results at screening:

   • ALT or AST > 2x the upper limit of the normal range
4. History of regular alcohol consumption exceeding 210 g/week within the 6 months prior to screening (1 drink (250 mL) of beer (5%) = 10 g; 1 drink (50 mL) of hard liquor (20%) = 8 g; 1 drink (125 mL) of wine (12%) = 12 g)
5. Individuals who smoked more than 20 cigarettes per day within 6 months prior to screening
6. Individuals who had been administered investigational product(s) from other clinical study or bioequivalence study within the 6 months prior to the first dose of this study
7. Following vital signs results at screening

   - Sitting systolic blood pressure ≥ 140 mmHg or < 90 mmHg and/or sitting diastolic blood pressure ≥90 mmHg or <60 mmHg
8. Individuals with a medical history of significant alcohol or drug abuse within one year prior to the screening
9. Individuals who had taken any drug(s) known as a strong inducer(s) or inhibitor(s) of drug-metabolizing enzymes within 30 days prior to the first dose of investigational product(s)
10. Individuals who had taken prescription or nonprescription drugs within the 10 days prior to the first dose of investigational product(s)
11. Individuals who donated whole blood within the 2 months, or blood components within 1 month prior to the first dose of the investigational product(s)
12. Individuals with severe acute/chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product(s) administration, or may interfere with the interpretation of study results
13. Individuals with hypersensitivity to investigational products or the investigational products ingredients or dihydropyridine drugs
14. Subject had severe heart failure(NYHA class 1, 2, 3, 4)
15. Patients with hepatopathy
16. Patients with diabetic ketogenic acidosis, diabetic comas and ex-coma, type 1 diabetes.
17. Before and after surgery, severe infections, severe trauma.
18. Patients with edema
19. Subject had renal impairment(eGFR < 60 mL/min/1.73 m²)
20. Subject who is a pregnant or nursing woman
21. Subject had genetic dysfunctions like galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
22. Subjects who were deemed inappropriate to participate in the study by the investigator

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-398 | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-dose
  Area under the plasma concentration time curve of CKD-344, from time zero up to the last measurable concentration.
Cmax of CKD-398 | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-dose
  The maximum concentration observed of CKD-344 over blood sampling time.

SECONDARY OUTCOMES:
AUCinf of CKD-398 | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-dose
  Area under the concentration-time curve from zero up to ∞
Tmax of CKD-398 | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-dose
  Time to maximum plasma concentration
T1/2 of CKD-398 | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-dose
  Terminal elimination half-life
CL/F of CKD-398 | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-dose
  Apparent Clearance
Vd/F of CKD-398 | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours post-dose
  Apparent volume of distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No